CLINICAL TRIAL: NCT01381744
Title: A Phase I Safety and Immunogenicity Dose Escalation Trial of Plague Vaccine, Flagellin/F1/V, In Healthy Adult Volunteers
Brief Title: Dose Escalation Trial of a Plague Vaccine, Flagellin/F1/V, in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 08-0066; Parent Protocol of 15-0104
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2014-10

CONDITIONS: Plague
Keywords: Yersinia pestis, vaccine, plague, Flagellin/F1/V, Parent Protocol of 15-0104
MeSH Terms: conditions — Plague

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group 3: 6 mcg Flagellin/F1/V (Experimental): 12 subjects will receive 6 mcg of Flagellin/F1/V or placebo on Day 0 and Day 28.
  Interventions: Biological: Flagellin/F1/V; Other: Placebo
- Group 4: 10 mcg Flagellin/F1V (Experimental): 12 subjects will receive 10 mcg of Flagellin/F1/V or placebo on Day 0 and Day 28.
  Interventions: Biological: Flagellin/F1/V; Other: Placebo
- Group 2: 3 mcg Flagellin/F1/V (Experimental): 12 subjects will receive 3 mcg of Flagellin/F1/V or placebo on Day 0 and Day 28.
  Interventions: Biological: Flagellin/F1/V; Other: Placebo
- Group 1: 1 mcg Flagellin/F1/V (Experimental): 12 subjects will receive 1 microgram (mcg) of Flagellin/F1/V or placebo on Day 0 and Day 28.
  Interventions: Biological: Flagellin/F1/V; Other: Placebo

INTERVENTIONS:
Biological: Flagellin/F1/V — Flagellin/F1/V recombinant fusion protein vaccine administered by the intramuscular route on Days 0 and 28 at a dose of 1, 3, 6, or 10 micrograms (mcg). It is a clear, colorless solution.
Other: Placebo — Phosphate buffered saline (PBS) used as diluent and placebo.

SUMMARY:
Plague is an infectious disease of animals and humans caused by bacteria, Yersinia pestis. Modern antibiotics are effective against plague, but if an infected person is not treated promptly the disease is likely to cause illness or death. The purpose of this study is to evaluate at the safety, immunogenicity (bodily defense reaction), and tolerability of a new research vaccine. Up to 48 people will be enrolled in this study at the Center for Vaccine Development at Saint Louis University. Four groups of 12 volunteers will be given vaccine or placebo (inactive substance) one group at a time starting with the lowest dose working up to the highest dose. Shots will be given in the arm 2 times separated by 28 days. Study procedures include: physical exam, blood samples, and recording temperature and side effects in a memory aid. Participants will be involved in study related procedures for about 13 months.

DETAILED DESCRIPTION:
Yersinia (Y.) pestis, a gram-negative coccobacillus, causes an acute and often fatal disease that may appear in 1 of several major manifestations: bubonic, septicemic, and pneumonic. Transmission to humans most commonly occurs via a bite by infectious fleas and is associated with regional lymphadenopathy or bubo. Pneumonic plague would be the most likely outcome in the case of a bio-terrorism attack. Currently, there is no effective licensed vaccine that protects against pneumonic plague. The investigational product, flagellin/F1/V in phosphate-buffered saline, pH 6.2, is a vaccine that is designed to provide protection against respiratory exposure to Y. pestis, i.e., pneumonic plague. The general hypothesis to be tested is that the flagellin/F1/V vaccine will induce a robust humoral immune response against the F1 and V antigens of Y. pestis without serious adverse events (SAEs) when the vaccine is given intramuscularly (IM) on 2 occasions separated by about 28 days at doses of 1, 3, 6 and 10 micrograms (mcg). Since the major rationale for this vaccine is protection against respiratory exposure to Y. pestis following a bio-terrorism attack, the initial study population will be 18-45 year old healthy volunteers. The primary objective of this study is to assess the safety and immunogenicity of escalating dosages of Flagellin/F1/V vaccine among healthy subjects given 2 doses of vaccine by the IM route on Days 0 and 28. The secondary objective of this study is to evaluate the reactogenicity and cell mediated immune responses of escalating dosages of Flagellin/F1/V vaccine among healthy subjects when given 2 doses of vaccine by the IM route on Days 0 and 28. Participants will include up to 48 healthy male and female volunteers. This study is designed as a randomized, placebo controlled, double-blind (within dosing group), dose escalation Phase I study. The study will consist of 4 groups to be dosed sequentially. Each group will consist of 10 individuals that receive vaccine and 2 that receive placebo. Each subject will receive an IM vaccination on Days 0 and 28. The initial dose to be evaluated will be 1 mcg/dose. Following assessment of safety and reactogenicity data of each group by the Safety Monitoring Committee the vaccine doses will be increased sequentially from 1, to 3, to 6, to 10 mcg/dose. Following vaccination, subjects will return to the clinical site on Days 1, 14, and 28 following the initial vaccination and on Days 1, 14, 28, 40, and 180 following the second vaccination. In addition, subjects will be contacted by phone on Day 3 after each vaccination to review the memory aid, query for adverse event (AEs)/SAEs and concomitant medications. All subjects will complete a subject memory aid for 15 days following each vaccination (Day 0-14). Unsolicited, non-serious AEs will be collected through Day 56 (Visit 8, 26-30 days following the final vaccination). SAEs will be collected throughout the study period Day 393 (Visit 11, 365 days + 14 days after the second vaccination). Blood samples for safety labs will be collected at screening, day of initial vaccination and at 14 days after each vaccination. Specimens will be collected for immunologic assays at the noted clinic visits, as well as at 6 months post the final vaccination.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria that must met prior to the initial vaccination:

* At least 18 and less than or equal to 45 years of age at the time of first vaccination.
* Never had plague or disease caused by Yersinia pestis.
* Able to provide informed consent.
* Read, signed, and dated informed consent document.
* Available for follow-up for the planned duration of the study.
* Satisfactory medical assessment with no clinically significant and relevant abnormalities as established by medical history and physical examination at screening.
* If the subject is female and of childbearing potential, negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to each vaccination.
* If the subject is female and of childbearing potential, she agrees to use acceptable contraception and remain on the same method during the study as they were using prior to entering the study, and not become pregnant for 28 days following the last vaccination. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. Acceptable contraception methods are restricted to effective devices [e.g., intrauterine device (IUD), NuvaRing®] or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, a monogamous relationship with a vasectomized partner and abstinence from sexual intercourse with men.
* Negative enzyme-linked immunosorbent assay (ELISA) for human immunodeficiency virus (HIV).
* Negative hepatitis B surface antigen and negative antibody to hepatitis C virus.
* Safety labs have to be within institutional normal limits, or as otherwise specified.
* Weight: greater than or equal to 110 pounds.
* Body Mass Index (BMI) of greater than or equal to 19 and less than 33.
* Subject agrees not to donate blood for the duration of their study participation.

Inclusion criteria that must be met prior to the second vaccination:

* Never had plague or disease caused by Yersinia pestis.
* Satisfactory medical assessment with no clinically significant and relevant abnormalities as established by medical history.
* If the subject is female and of childbearing potential, negative urine or serum pregnancy test within 24 hours prior to vaccination.
* If the subject is female and of childbearing potential, she has remained on the same contraception method as used prior to entering the study, and not become pregnant for 28 days following the last vaccination. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. Acceptable contraception methods are restricted to effective devices (e.g., IUDs, NuvaRing®) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, a monogamous relationship with a vasectomized partner and abstinence from sexual intercourse with men.
* Post dose one safety labs (Day 14) have to be within institutional normal limits, or as otherwise specified at the Day 14 post the initial vaccination or any observed laboratory toxicities have to be resolved prior to the second vaccination.

Exclusion Criteria:

Exclusion criteria prior to 1st vaccination:

* History of immunodeficiency or suspected impairment of immunologic functioning.
* Known or suspected history of plague vaccination.
* Pregnant women or women that are breastfeeding.
* Uncontrolled hypertension (defined as systolic blood pressure >140 mm Hg and/or diastolic blood pressure > 90 mm Hg).
* Subject is on statin therapy.
* 10% or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hin.nhlbi.nih.gov/atpiii/calculator.asp). NOTE that this criterion applies only to subjects 20 years of age and older AND only if at least one of the following apply: have smoked a cigarette in the past month, have hypertension (defined as systolic blood pressure >140 mm Hg) or are on antihypertensive medication and/or have a family history of coronary heart disease in male first-degree relative (father or brother) <55 years of age or a female first-degree relative (mother or sister) <65 years of age.
* Current use or use within 30 days of screening of immunosuppressive medication or corticosteroids (use of topical or nasal corticosteroids is allowed). Persons who are using a topical steroid can be enrolled after their therapy is completed. Inhaled steroids for asthma are not permissible.
* Chronic use of non-steroidal anti-inflammatory drug therapy
* Malignancy not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site or history of skin cancer at the vaccination site.
* Active autoimmune disease [Persons with vitiligo or thyroid disease (e.g., taking thyroid hormone replacement) are not excluded].
* Receipt of any vaccine 14 days prior to vaccination.
* Receipt of live attenuated vaccine within 30 days prior to vaccination.
* Planned receipt of any vaccine including allergy shots during the 28 day vaccination period and through 14-days post the second vaccination (Visit 7).
* Receipt of blood products or immunoglobulin within six months prior to vaccination.
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol.
* Use of any other experimental agent (i.e. chemical or biological entity not registered for clinical use) within 30 days prior to vaccination and for the duration of the study
* Donation of a unit of blood within 56 days prior to vaccination.
* Acute febrile illness (>100.2 degrees F) on the day of vaccination.
* Any condition that, in the opinion of the investigator, might interfere with study objectives or would make administration of the study vaccine hazardous or make it difficult to monitor adverse effects.
* Study personnel.
* Current abuse of alcohol or drug addiction that in the opinion of the Investigator may interfere with the subject's ability to comply with trial procedures.

Exclusion criteria that apply prior to second vaccination:

* Subject that were discontinued due to meeting individual halting rule after the first vaccination.
* History of immunodeficiency or suspected impairment of immunologic functioning.
* Known or suspected history of plague vaccination, excluding the vaccine received as part of this study.
* Pregnant women or women that are breastfeeding.
* Uncontrolled hypertension (defined as systolic blood pressure >140 mm Hg and/or diastolic blood pressure > 90 mm Hg).
* Subject is on statin therapy
* Current use or use since initial vaccination of immunosuppressive medication or corticosteroids (use of topical or nasal corticosteroids is allowed). Persons who are using a topical steroid can be enrolled after their therapy is completed. Inhaled steroids for asthma are not permissible.
* Malignancy not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site or history of skin cancer at the vaccination site.
* Active autoimmune disease [Persons with vitiligo or thyroid disease (e.g., taking thyroid hormone replacement) are not excluded].
* Receipt of any vaccine 14 days prior to vaccination.
* Receipt of live attenuated vaccine within 30 days prior to vaccination.
* Receipt of blood products or immunoglobulin since initial vaccination.
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol.
* Use of any other experimental agent (i.e. chemical or biological entity not registered for clinical use) within 30 days prior to vaccination and for the duration of the study.
* Donation of a unit of blood within 56 days prior to vaccination.
* Subject experienced a Grade 2 or higher fever (equal or greater than 101.6 °F) within the first 24 hours following the initial study vaccination.
* Acute febrile illness (>/= 100.0 °F) on the day of vaccination.
* Any condition that, in the opinion of the investigator, might interfere with study objectives or would make administration of the study vaccine hazardous or make it difficult to monitor adverse effects.
* Study personnel.
* Current abuse of alcohol or drug addiction that in the opinion of the Investigator may interfere with the subject's ability to comply with trial procedures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade 3 or above laboratory toxicities associated with vaccination for each dose group. | Through Day 42 (14 days after the second vaccination).
Incidence of serious adverse events (SAEs)associated with vaccination for each dose group. | Throughout the duration of the study (Visit 11, 365 + 14 days after the second vaccination or through termination visit, if terminated early).
Peak antibody titer [immunoglobulin G (IgG) enzyme-linked immunosorbent assay (ELISA) for F1 and V antigen] for each dose group as determined by analysis of serum samples. | Days: 0, 14, 28, 42, 56, 68 and 208.

SECONDARY OUTCOMES:
Distribution of the cytokine expression levels in peripheral blood mononuclear cells (PBMCs) following ex vivo stimulation for each dose group. | Day 0, 14, 42, 56, and 68.
Occurrence of unsolicited adverse events (AEs) for each dose group. | Within 28 days of each vaccination.
Occurrence of systemic reactogenicity symptoms for each dose group. | Within 15 days (Day 0-14) of each vaccination.
Occurrence of localized reactogenicity symptoms for each dose group. | Within 15 days (Day 0-14) of each vaccination.
Assessment of cytokine responses (TNF-alpha, IL-6 and IL-1 beta) as measured in serum samples. | Serum samples obtained on the day of vaccination, and on Visit 3 and 6 (1 day after each vaccination) and Visit 4 and 7 (14 days after each vaccination).

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University - Center for Vaccine Development, St Louis, Missouri, United States